CLINICAL TRIAL: NCT00113867
Title: Effects of Hormonal Infertility Treatment on Cognition in Pre-Menopausal Women
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Other Study IDs: AG0022
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2006-11

CONDITIONS: Infertility
Keywords: IVF; in vitro fertilization; hormones; stress; memory; Cognitive Function; adoption
MeSH Terms: conditions — Infertility

SUMMARY:
The purpose of this study is to examine the effects of marked alterations in ovarian steroid hormones on cognitive functions in women. Sex hormones and stress hormones of women awaiting or undergoing in-vitro fertilization (IVF) will be compared with levels of women adopting children and women on oral contraceptives.

DETAILED DESCRIPTION:
Much of our understanding of the effects of ovarian steroid hormones on cognitive functioning comes from studies of changes in cognitive function associated with hormone replacement therapy (HRT) in post-menopausal women and changes in menstrual cycle phase in premenopausal women. If fluctuations in ovarian sex steroid hormone levels across the normal physiological range affect cognitive functions in women, then marked alterations in hormone levels should have a notable effect on cognitive function.

Hormonal in-vitro fertilization (IVF) treatments for female infertility result in dramatic fluctuations in estrogen levels. Women awaiting infertility treatment report negative emotions, depressed mood, declines in memory and concentration, and higher levels of reported stress compared to women who have never experienced infertility.

Four groups of twenty women each will be recruited for this observational study:

* Group 1 - IVF treatment with GnRH-a alone
* Group 2 - IVF treatment with GnRH-a plus sex steroid stimulating hormones
* Group 3 - ADPT control (women in the process of adopting children)
* Group 4 - OC (oral contraceptives) control

All groups will receive a cognitive/affect assessment twice, with a 3-week interval between assessments. Blood and salivary samples will be taken on the two test days to measure ovarian sex steroid hormone levels and stress hormone levels. Salivary samples will also be taken on a third day in between the two test days. Heart Period Variability (HPV), a measure of cardiac functioning, will be measured using electrocardiogram (ECG).

ELIGIBILITY:
Inclusion Criteria:

* Women 25 years and older, who are still ovulating
* Residing in Maryland or the Washington DC metropolitan area
* Healthy women in one of the following groups:
* 1) beginning or currently undergoing IVF infertility treatments with GnRH-a alone,
* 2) beginning or currently undergoing IVF infertility treatments with GnrH-a plus sex steroid stimulating hormones,
* 3) going through the adoption process, or
* 4) taking monophasic oral contraceptives for at least six months

Exclusion Criteria:

* English not the primary language
* Women who are peri- or post-menopausal
* Women who are currently taking anti-depressants or have a history of head injury or neurological/psychiatric condition
* Groups 1 & 2 (IVF) - women who are undergoing Inter-uterine insemination as an infertility treatment
* Group 3 (ADPT) - women who underwent hormonal infertility treatments within the previous 6 months
* Group 4 (OC) - women on progesterone only (mini-pill) oral contraceptives

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2003-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa H. Kitner-Triolo, PhD, Principal Investigator — Research Psychologist, Laboratory of Personality & Cognition, Cognition Section, Intramural Reserach Program, National Institute on Aging, National Institutes of Health
Locations (1):
- National Institute on Aging (NIA), Harbor Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Sherwin BB, Tulandi T. "Add-back" estrogen reverses cognitive deficits induced by a gonadotropin-releasing hormone agonist in women with leiomyomata uteri. J Clin Endocrinol Metab. 1996 Jul;81(7):2545-9. doi: 10.1210/jcem.81.7.8675575.
- [Background] Harlow CR, Fahy UM, Talbot WM, Wardle PG, Hull MG. Stress and stress-related hormones during in-vitro fertilization treatment. Hum Reprod. 1996 Feb;11(2):274-9. doi: 10.1093/humrep/11.2.274. PMID 8671208
- [Background] Oddens BJ, den Tonkelaar I, Nieuwenhuyse H. Psychosocial experiences in women facing fertility problems--a comparative survey. Hum Reprod. 1999 Jan;14(1):255-61. doi: 10.1093/humrep/14.1.255. PMID 10374131